CLINICAL TRIAL: NCT03863574
Title: A Phase 2, Prospective, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Saroglitazar Magnesium 2 mg and 4 mg in Patients With Non-alcoholic Steatohepatitis (NASH)
Brief Title: Saroglitazar Magnesium in the Treatment of Non-Alcoholic Steatohepatitis
Acronym: EVIDENCES VI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SARO.17.004
Record Dates: First submitted 2019-02-24; First posted 2019-03-05 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Non Alcoholic Steatohepatitis
Keywords: NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — saroglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Saroglitazar Magnesium 2 mg (Experimental): Saroglitazar Magnesium 2 mg tablet orally once daily in the morning before breakfast for 24 weeks.
  Interventions: Drug: Saroglitazar Magnesium 2mg
- Saroglitazar Magnesium 4 mg (Experimental): Saroglitazar Magnesium 4 mg tablet orally once daily in the morning before breakfast for 24 weeks.
  Interventions: Drug: Saroglitazar Magnesium 4mg
- Placebo (Placebo Comparator): Placebo tablet orally once daily in the morning before breakfast for 24 weeks.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Saroglitazar Magnesium 2mg — Patients randomly assigned to this group will receive Saroglitazar Magnesium 2 mg tablet orally once daily for 24 weeks.
  Arms: Saroglitazar Magnesium 2 mg
Drug: Saroglitazar Magnesium 4mg — Patients randomly assigned to this group will receive Saroglitazar Magnesium 4 mg tablet orally once daily for 24 weeks.
  Arms: Saroglitazar Magnesium 4 mg
Drug: Placebos — Patients randomly assigned to this group will receive Placebo tablet orally once daily for 24 weeks.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to evaluate safety and efficacy of Saroglitazar Magnesium 2 mg and 4 mg in patients with NASH. This study will be initiated after obtaining the approvals of Institutional Ethics Committee/Institutional Review Board (IEC/IRB) and the local regulatory authority.

DETAILED DESCRIPTION:
Patients clinically suspected of NASH will be invited for a screening programme for inclusion in the study. Patients will be screened according to the inclusion and exclusion criteria. Clinical evaluation will be conducted for baseline characteristics and anthropometry measurements such as body weight and height.

After clinical evaluations, all baseline safety and efficacy parameters will be recorded as per Visit Schedule. All laboratory collections will be performed following overnight fasting (at least 8 hrs).

Following confirmation of all clinical and laboratory inclusion and exclusion criteria, patients will continue into the screening period. During the screening period liver biopsy will be performed. However, if a biopsy was performed within 6 months the slides and biopsy material, or block, must be made available for baseline documentation. Such Patients, whose historical biopsy report is available, should not use medication suspected of having an effect on NASH from the 3 months prior to the screening.

Liver biopsy will be performed to confirm the diagnosis of NASH and record a baseline Non-alcoholic fatty liver disease (NAFLD) Activity Score (NAS). The histological evidence of NASH is defined as NAS ≥ 4 with a minimum score of 1 for all of its three components [steatosis, hepatocyte ballooning and lobular inflammation].

Following confirmation of inclusion/exclusion criteria and upon histological confirmation of NASH by liver biopsy, patients will be enrolled into the study.

Eligible patients will be randomly assigned to receive Saroglitazar Magnesium 2 mg or 4 mg or placebo in a 2:2:1 ratio for 24 weeks.

Upon completion of 24 weeks of treatment, liver biopsy will be performed and the NAFLD Activity Score recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to provide written informed consent for participation in this trial.
2. Males or females, 18 to 75 years of age, both inclusive.
3. Female must be either of non-child bearing potential (surgically sterilized at least 6 months prior to screening or postmenopausal) or using one or more methods of contraception.
4. Histologic confirmation of NASH without cirrhosis (fibrosis stage 0, 1, 2, or 3) from liver biopsy performed either during the screening period or no more than 6 months prior to the first visit, with a NAS of ≥4 and a score of at least 1 in each (steatosis scored 0-3, ballooning scored 0-2, and lobular inflammation scored 0-3). If biopsy was performed within 6 months of screening, the slides, biopsy material or block should be available for baseline documentation. Such patients, whose historical biopsy report is available, should not use medications suspected of having an effect on NASH for at least 3 months prior to the screening.
5. BMI ≥25 kg/m^2.
6. For hypertensive patients, blood pressure must be controlled by a stable dose of antihypertensive medications for at least 3 months prior to screening (and the stable dose can be maintained throughout the study)
7. Patients with type 2 diabetes mellitus may be included if they fulfil the following criteria;

   1. Stable therapeutic regimen as defined by no changes in oral agents or dose for at least 3 months before screening and the stable dose can be maintained throughout the study.
   2. HbA1c ≤ 9.5%
8. Patients agree to comply with the study procedure.

Exclusion Criteria:

1. Pregnant and lactating female.
2. Positive pregnancy test.
3. Patients with history of myopathies or evidence of active muscle diseases.
4. Patients with history of alcohol consumption of >30 gm/day for men, >20 gm/day for women for consecutive previous 2 years and/or drug abuse.
5. Known allergy, sensitivity or intolerance to the study drug or formulation ingredients.
6. Participation in an interventional clinical study and/or receipt of any investigational medication within 3 months prior to screening.
7. History of malignancy in the past 5 years and/or active neoplasm with the exception of superficial, non-melanoma, skin cancer.
8. Any of the following laboratory values at screening:

   1. Direct bilirubin >1.5 mg/dL,
   2. Serum albumin <2.5 g/dL.
   3. Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m2.
   4. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >200 IU/L.
   5. Patient with international normalized ratio (INR) >1.5.
   6. Creatinine kinase ≥ 1.5 upper limit of normal (ULN).
   7. Lipase ≥ULN.
   8. Amylase ≥ ULN.
9. Unstable cardiovascular disease, including:

   1. unstable angina, (i.e., new or worsening symptoms of coronary heart disease within the 3 months preceding screening), acute coronary syndrome within the 6 months preceding Screening, acute myocardial infarction within the 3 months preceding screening or heart failure of New York Heart Association class (III - IV) or worsening congestive heart failure, or coronary artery intervention, within the 6 months preceding screening
   2. history of (within 3 months preceding Screening) or current unstable cardiac dysrhythmias
   3. uncontrolled hypertension (systolic blood pressure [BP] > 155 mmHg and/or diastolic BP > 95 mmHg)
   4. Stroke or transient ischemic attack within the 6 months preceding screening.
10. Previous history of bladder disease and/or hematuria.
11. Previous liver biopsy that demonstrated presence of cirrhosis or radiologic imaging consistent with cirrhosis or portal hypertension.
12. Type 1 diabetes mellitus.
13. Use of drugs that are known Cytochrome P4502C8 (CYP2C8) inhibitors/substrate.
14. Use of drugs associated with a clinical or histological picture consistent with fatty liver disease or NASH for more than 12 consecutive weeks in the 1 year prior to start of the study; (these include amiodarone, tamoxifen, methotrexate, glucocorticoids, anabolic steroids, tetracyclines, estrogens, valproate/valproic acid, chloroquine, anti-HIV drugs).
15. History of thyroid disease (hypothyroid patients who are euthyroid on thyroid hormone replacement can be included).
16. History of, or current, cardiac dysrhythmias.
17. History of bariatric surgery, or undergoing evaluation for bariatric surgery.
18. Patients with a >10% weight loss in the 3 months prior to screening.
19. History or other evidence of severe illness or any other conditions that would make the patient, in the opinion of the Investigator, unsuitable for the study (such as poorly controlled psychiatric disease, coronary artery disease, HIV or active gastrointestinal conditions that might interfere with drug absorption).
20. Patients on any treatment with other drugs used for treatment of NASH [pentoxyphyllin, ursodeoxycholic acid, antioxidants such as vitamin E (>800 IU/day), glutathione, orlistat, betaine, incretin mimetics or non-prescribed complementary alternative medications (including dietary supplements, megadose vitamins, herbal preparations and special teas)] or any medicine in clinical trials for NASH. (However, patients who are taking stable dose of vitamin E for at least 3 months prior to screening will be enrolled in the study).
21. History of other causes of chronic liver disease [autoimmune, primary biliary cirrhosis, hepatitis B virus (HBV) and hepatitis C virus (HCV), Wilson disease, alpha-1-antitrypsin deficiency, hemochromatosis etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deven V Parmar, MD,FACP,FCP, Study Director — Zydus Therapeutics Inc.
Locations (6):
- United States (6):
  - Southern Therapy and Advanced Research (STAR) LLC, Jackson, Mississippi
  - Gastro One, Germantown, Tennessee
  - Digestive Health Research, Hermitage, Tennessee
  - Texas Liver Institute, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Background] Siddiqui MS, Parmar D, Sheikh F, Sarin SK, Cisneros L, Gawrieh S, Momin T, Duseja A, Sanyal AJ. Saroglitazar, a Dual PPAR alpha/gamma Agonist, Improves Atherogenic Dyslipidemia in Patients With Non-Cirrhotic Nonalcoholic Fatty Liver Disease: A Pooled Analysis. Clin Gastroenterol Hepatol. 2023 Sep;21(10):2597-2605.e2. doi: 10.1016/j.cgh.2023.01.018. Epub 2023 Jan 31. PMID 36731585
- [Result] Siddiqui MS, Idowu MO, Parmar D, Borg BB, Denham D, Loo NM, Lazas D, Younes Z, Sanyal AJ. A Phase 2 Double Blinded, Randomized Controlled Trial of Saroglitazar in Patients With Nonalcoholic Steatohepatitis. Clin Gastroenterol Hepatol. 2021 Dec;19(12):2670-2672. doi: 10.1016/j.cgh.2020.10.051. Epub 2020 Nov 2. PMID 33152542
- See also: Siddiqui MS, Parmar D. Saroglitazar, a Dual PPAR alpha/gamma Agonist, Improves Atherogenic Dyslipidemia in Patients With Non-Cirrhotic Nonalcoholic Fatty Liver Disease: A Pooled Anal — http://pubmed.ncbi.nlm.nih.gov/36731585/
- See also: Siddiqui MS, Idowu MO, Parmar D, Borg BB, Denham D, Loo NM, Lazas D, Younes Z, Sanyal AJ. A Phase 2 Double Blinded, Randomized Controlled Trial of Saroglitazar in Patients With Nonalcoholic Steatohepatitis — http://pubmed.ncbi.nlm.nih.gov/33152542/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Started | 6 | 7 | 3
Completed | 6 | 7 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 3 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.67 (9.91) | 50.57 (16.48) | 63.33 (8.08) | 52.25 (13.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 14
  Male | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 1 | 5
  Not Hispanic or Latino | 5 | 3 | 2 | 10
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 5 | 7 | 2 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 7 | 3 | 16
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 37.32 (5.85) | 37.89 (8.27) | 37.67 (12.76) | 37.63 (7.78)

OUTCOME MEASURES:

1. Primary Outcome: NAS Score (Nonalcoholic Fatty Liver Disease [NAFLD] Activity Score)
Description: The primary endpoint is to assess the changes in NAFLD Activity Score (NAS) at week 24 from baseline and with no worsening of fibrosis in NASH patients.
  NAFLD Activity Score Steatosis <5% - 0 5% -33% - 1 >33% -66% - 2 >66% - 3 Lobular Inflammation No foci - 0 <2 foci per 200 X field -1 2-4 foci per 200 X field - 2 >4 foci per 200 X field - 3 Ballooning None - 0 Few balloon cells -1 Many cells/prominent ballooning - 2 Final NAFLD Activity Score = Steatosis Score + Lobular Inflammation Score + Ballooning Score Minimum score for NAS is 0 Maximum score for NAS is 8 Higher score represents the worse disease activity
Time Frame: Baseline to Week 24
Population: modified intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
units on a scale | -1.50 (0.84) | -1.86 (1.57) | -1.33 (0.58)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof of Concept; p = 0.7689, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.6007, t-test, 2 sided

2. Secondary Outcome: To Evaluate the Percentage of Responders in the Treatment Groups.
Description: Responder is defined as a decrease from baseline of at least 2 points spread across at least 2 of the NAS components [steatosis, hepatocyte ballooning, and lobular inflammation] with no worsening of fibrosis.
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
Participants | 4 | 3 | 1
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other; p = 0.5238, Fisher Exact
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other; p > 0.9999, Fisher Exact

3. Secondary Outcome: Percentage of Responders Defined by the Disappearance of Steatohepatitis.
Description: Percentage of responders defined by the disappearance of steatohepatitis
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
Participants | 5 | 6 | 0
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.0476, Fisher Exact
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.0333, Fisher Exact

4. Secondary Outcome: Changes in the Stage of Steatosis, Lobular Inflammation and Ballooning.
Description: Changes in the stage of steatosis, lobular inflammation and ballooning by evaluating the NAS Score (Nonalcoholic fatty liver disease Activity Score)
  Steatosis <5% - 0 5% -33% - 1 >33% -66% - 2 >66% - 3 Lobular Inflammation No foci - 0 <2 foci per 200 X field -1 2-4 foci per 200 X field - 2 >4 foci per 200 X field - 3 Ballooning None - 0 Few balloon cells -1 Many cells/prominent ballooning - 2 Higher score represents the worse disease activity
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
units on a scale
  Changes in the stage of steatosis | -0.50 (0.55) | -0.71 (0.76) | -0.33 (0.58)
  Changes in the stage of lobular inflammation | -0.17 (0.41) | -0.29 (0.49) | -0.67 (0.58)
  Changes in the stage of ballooning | -0.83 (0.41) | -0.86 (0.90) | -0.33 (0.58)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Steatosis; Test type: Other — Proof-of-concept; p = 0.6845, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Steatosis; Test type: Other — Proof-of-concept; p = 0.4625, t-test, 2 sided
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Lobular Inflammation; Test type: Other — Proof-of-concept; p = 0.1705, t-test, 2 sided
Statistical Analysis 4: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome variable: Lobular Inflammation; Test type: Other — Proof-of-concept; p = 0.3122, t-test, 2 sided
Statistical Analysis 5: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Hepatocyte Ballooning; Test type: Other — Proof-of-concept; p = 0.1705, t-test, 2 sided
Statistical Analysis 6: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Hepatocyte Ballooning; Test type: Other — Proof-of-concept; p = 0.3877, t-test, 2 sided

5. Secondary Outcome: Changes in the Stage of Fibrosis.
Description: Changes in the stage of fibrosis by evaluating the Fibrosis stages
  Fibrosis Score
  Definition None - 0 Perisinusoidal or periportal - 1 Mild, zone 3, perisinusoidal - 1A Moderate, zone3, perisinusoidal -1B Portal/periportal -1C Perisinusoidal and portal/periportal - 2 Bridging fibrosis - 3 Cirrhosis - 4 Higher score represents the worse disease activity
Time Frame: Baseline to Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
units on a scale | -0.50 (0.84) | -0.43 (0.79) | 0.33 (0.58)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.1705, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.1740, t-test, 2 sided

6. Secondary Outcome: Changes in the Liver Function Tests; (Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST], Alkaline Phosphatases [ALP], and Gamma-glutamyl Transferase [GGT]).
Description: Liver function tests include ALT, AST, ALP, GGT
Time Frame: Baseline to Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
U/L
  Change in ALT | -22.83 (14.29) | -29.57 (26.76) | -14.67 (48.95)
  Change in AST | -10.33 (5.32) | -16.29 (11.63) | -19.33 (47.44)
  Change in ALP | -24.00 (9.92) | -23.86 (15.18) | 3.67 (5.13)
  Change in GGT | -23.83 (18.55) | -28.43 (33.30) | -1.67 (19.50)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome variable: Alanine Aminotransferase; Test type: Other — Proof-of-concept; p = 0.8019, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Alanine Aminotransferase; Test type: Other — Proof-of-concept; p = 0.5396, t-test, 2 sided
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Aspartate Aminotransferase; Test type: Other — Proof-of-concept; p = 0.7740, t-test, 2 sided
Statistical Analysis 4: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Aspartate Aminotransferase; Test type: Other — Proof-of-concept; p = 0.9221, t-test, 2 sided
Statistical Analysis 5: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Alkaline Phosphatase; Test type: Other — Proof-of-concept; p = 0.0030, t-test, 2 sided
Statistical Analysis 6: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Alkaline Phosphatase; Test type: Other — Proof-of-concept; p = 0.0177, t-test, 2 sided
Statistical Analysis 7: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Gamma Glutamyl Transferase; Test type: Other — Proof-of-concept; p = 0.1399, t-test, 2 sided
Statistical Analysis 8: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Gamma Glutamyl Transferase; Test type: Other — Proof-of-concept; p = 0.2384, t-test, 2 sided

7. Secondary Outcome: Changes in the Liver Function Tests; Albumin and Total Protein
Description: Changes in albumin and total protein
Time Frame: Baseline to Week 24
Population: Modified intend-to-treat population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
g/dL
  Change in albumin | -0.05 (0.22) | -0.04 (0.17) | 0.13 (0.12)
  Change in total protein | -0.08 (0.40) | 0.09 (0.41) | 0.27 (0.06)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Albumin; Test type: Other — Proof-of-concept; p = 0.2218, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Albumin; Test type: Other — Proof-of-Concept; p = 0.1483, t-test, 2 sided
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Total Protein; Test type: Other — Proof-of-concept; p = 0.0839, t-test, 2 sided
Statistical Analysis 4: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Total Protein; Test type: Other — Proof-of-concept; p = 0.2895, t-test, 2 sided

8. Secondary Outcome: Changes in the Liver Function Tests; Direct Bilirubin
Description: Change in direct bilirubin
Time Frame: Baseline to Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
mg/dL | -0.01 (0.03) | -0.01 (0.02) | -0.00 (0.02)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Direct Bilirubin; Test type: Other — Proof-of-concept; p = 0.6808, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Direct Bilirubin; Test type: Other — Proof-of-concept; p = 0.5351, t-test, 2 sided

9. Secondary Outcome: Changes in the Lipid Profile.
Description: Evaluation of Lipid profile parameters
Time Frame: Baseline to Week 24
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
mg/dL
  Change in Triglyceride | -40.33 (38.37) | -16.71 (44.31) | -6.00 (34.04)
  Change in Total Cholesterol | 11.17 (40.45) | -16.00 (31.12) | -0.33 (9.02)
  Change in Small dense LDL | 1.27 (15.99) | -9.29 (11.85) | 5.87 (6.66)
  Change in High-density Lipoprotein | 6.33 (14.85) | -0.14 (8.47) | 7.00 (4.36)
  Change in Low-density lipoprotein | 13.00 (34.89) | -12.57 (28.11) | -6.00 (5.29)
  Change in Very low-density lipoprotein | -8.17 (7.41) | -3.29 (8.88) | -1.33 (6.51)
  Change in non-HDL Cholesterol | 4.83 (33.68) | -15.86 (29.23) | -7.33 (9.29)
  Change in Apo lipoprotein A1 | 10.50 (36.74) | -14.29 (26.98) | 7.33 (2.08)
  Change in Apo lipoprotein B | 1.00 (26.53) | -14.71 (21.04) | -1.33 (4.62)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Triglyceride; Test type: Other — Proof-of-concept; p = 0.2329, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Triglyceride; Test type: Other — Proof-of-concept; p = 0.7211, t-test, 2 sided
Statistical Analysis 3: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variables: Total Cholesterol; Test type: Other — Proof-of-concept; p = 0.6520, t-test, 2 sided
Statistical Analysis 4: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Total Cholesterol; Test type: Other — Proof-of-concept; p = 0.4302, t-test, 2 sided
Statistical Analysis 5: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: High-density Lipoprotein; Test type: Other — Proof-of-concept; p = 0.9432, t-test, 2 sided
Statistical Analysis 6: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: High-density Lipoprotein; Test type: Other — Proof-of-concept; p = 0.2133, t-test, 2 sided
Statistical Analysis 7: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Low-density lipoprotein; Test type: Other — Proof-of-concept; p = 0.2446, t-test, 2 sided
Statistical Analysis 8: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Low-density lipoprotein; Test type: Other — Proof-of-concept; p = 0.7075, t-test, 2 sided
Statistical Analysis 9: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Very low-density lipoprotein; Test type: Other — Proof-of-concept; p = 0.2195, t-test, 2 sided
Statistical Analysis 10: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Very low-density lipoprotein; Test type: Other — Proof-of-concept; p = 0.7435, t-test, 2 sided
Statistical Analysis 11: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: non-HDL Cholesterol; Test type: Other — Proof-of-concept; p = 0.5702, t-test, 2 sided
Statistical Analysis 12: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: non-HDL Cholesterol; Test type: Other — Proof-of-concept; p = 0.6441, t-test, 2 sided
Statistical Analysis 13: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Apo lipoprotein A1; Test type: Other — Proof-of-concept; p = 0.8415, t-test, 2 sided
Statistical Analysis 14: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Apo lipoprotein A1; Test type: Other — Proof-of-concept; p = 0.0786, t-test, 2 sided
Statistical Analysis 15: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Apo lipoprotein B; Test type: Other — Proof-of-concept; p = 0.8878, t-test, 2 sided
Statistical Analysis 16: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome variable: Apo lipoprotein B; Test type: Other — Proof-of-concept; p = 0.3219, t-test, 2 sided
Statistical Analysis 17: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Outcome Variable: Small dense LDL; Test type: Other — Proof-of-concept; p = 0.6557, t-test, 2 sided
Statistical Analysis 18: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Outcome Variable: Small dense LDL; Test type: Other — Proof-of-concept; p = 0.0763, t-test, 2 sided

10. Secondary Outcome: Number of Participants Experiencing Adverse Events After Consuming Saroglitazar Magnesium 2 mg and 4 mg
Description: Number of Participants with Adverse Events.
Time Frame: Baseline to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
Participants | 3 | 5 | 2

11. Secondary Outcome: Changes in the Glycemic Control and Insulin Resistance; Fasting Plasma Glucose
Description: Evaluation of Fasting Plasma Glucose
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
mg/dL | 2.67 (19.18) | -0.86 (41.10) | 7.67 (12.50)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.6988, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.7413, t-test, 2 sided

12. Secondary Outcome: Changes in the Glycemic Control and Insulin Resistance; Hemoglobin A1c
Description: Evaluation of Hemoglobin A1c
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
percentage of HbA1c | -0.52 (0.65) | -0.09 (0.28) | 0.03 (0.35)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.2200, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.5798, t-test, 2 sided

13. Secondary Outcome: Changes in the Glycemic Control and Insulin Resistance; Insulin
Description: Evaluation of Insulin
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
μIU/mL | -1.05 (20.05) | 6.74 (15.34) | 8.13 (12.32)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.4981, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.8939, t-test, 2 sided

14. Secondary Outcome: Changes in the Glycemic Control and Insulin Resistance: C-peptide
Description: Evaluation of C-peptide
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
ng/mL | -1.09 (2.26) | 0.08 (1.41) | 0.27 (0.95)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.3605, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.8394, t-test, 2 sided

15. Secondary Outcome: Changes in the Glycemic Control and Insulin Resistance: Homeostasis Model Assessment of Beta Cell Function (HOMA -β)
Description: Evaluation of HOMA of Beta Cell Function Homeostasis model assessment of beta cell function measures as following; HOMA -β = fasting insulin (μU/mL) ×360/{fasting glucose (mg/dL) - 63}.
  HOMA-B provides a quantitative estimate of beta-cell function. A lower HOMA-B value indicates reduced beta-cell function, which can be a sign of progressing towards or already having type 2 diabetes. Conversely, a higher HOMA-B value suggests better beta-cell functionality.
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percentage of HOMA of Beta Cell Function
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
percentage of HOMA of Beta Cell Function | -34.35 (84.41) | 14.49 (358.04) | 30.10 (46.15)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.2665, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.9133, t-test, 2 sided

16. Secondary Outcome: Changes in the Glycemic Control and Insulin Resistance: HOMA of Insulin Resistance
Description: Evaluation of HOMA of Insulin Resistance Insulin Resistance Index measures insulin resistance, calculated by fasting insulin (μU/mL) multiplied by fasting glucose (mg/dL), and divided by a constant (405). A higher score indicates higher insulin resistance.
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percentage of HOMA of Insulin Resistance
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
percentage of HOMA of Insulin Resistance | 0.45 (8.30) | 2.73 (5.77) | 2.34 (4.18)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.7267, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.9211, t-test, 2 sided

17. Secondary Outcome: Changes in the Glycemic Control and Insulin Resistance: Total Adiponectin
Description: Evaluation of Total Adiponectin
Time Frame: Baseline to Week 24
Population: modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
Number analyzed (Participants) | 6 | 7 | 3
μg/mL | 1.84 (2.17) | 0.68 (3.28) | 1.50 (4.02)
Statistical Analysis 1: Comparison: Saroglitazar Magnesium 2 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.8683, t-test, 2 sided
Statistical Analysis 2: Comparison: Saroglitazar Magnesium 4 mg vs Placebo; Test type: Other — Proof-of-concept; p = 0.7436, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Saroglitazar Magnesium 2 mg | Saroglitazar Magnesium 4 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 2/7 | 0/3
Other Adverse Events (participants affected / at risk) | 3/6 | 5/7 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saroglitazar Magnesium 2 mg (N=6) | Saroglitazar Magnesium 4 mg (N=7) | Placebo (N=3)
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saroglitazar Magnesium 2 mg (N=6) | Saroglitazar Magnesium 4 mg (N=7) | Placebo (N=3)
Influenza (Infections and infestations) | 0 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Uvulitis (Gastrointestinal disorders) | 0 | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Allergy to animal (Immune system disorders) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03863574/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT03863574/SAP_001.pdf